CLINICAL TRIAL: NCT01923324
Title: Physician to Physician Telephone Consultation for Chronic Pain Patients: a Pragmatic Randomized Trial
Brief Title: Standard Telephone Consultation for Pain
Acronym: STC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Project ID 18618
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician telephone consultation (Experimental): Received direct telephone consultation with pain physician about index patient
  Interventions: Behavioral: Physician telephone consultation
- Usual family physician care (Active Comparator): Usual family physician care (without direct telephone consultation with pain physician)
  Interventions: Behavioral: Usual family physician care

INTERVENTIONS:
Behavioral: Physician telephone consultation — Pain physician support for family physician treating patient
  Arms: Physician telephone consultation
Behavioral: Usual family physician care — Usual family physician care without telephone consultation with pain physician
  Arms: Usual family physician care

SUMMARY:
The purpose of this study is to investigate whether pain control for patients with chronic pain is improved by the availability of structured telephone consultations between the patients' family physicians and pain physicians, compared to pain control for patients receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to Alberta Health Services chronic pain center in Calgary with neurological or muscular skeletal pain

Exclusion Criteria:

* increased risk for suicide, very complex patients, family physician could not reliably identify patient's pain problem, or condition warranted expedited consultation with pain physician, case represented a new presentation of chronic regional pain syndrome, or low back pain with radicular symptoms or sciatica

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale for pain intensity (NRS) | 6 months
  11 point scale (from zero to 10), zero equals no pain, 10 worst possible pain.

SECONDARY OUTCOMES:
Pain Disability Index (PDI) | 6 months
  7 item self-report scale assessing pain disability
Patient Global Impression of Change Scale (PGIC) | 6 months
  7 point scale
Short Form Health Survey (SF-36) | 6 months
  Generic quality of life scale.

OTHER OUTCOMES:
Pain treatment satisfaction scale (patient) | 6 months
Family physician satisfaction questionnaire | 6 months
Family physician knowledge transfer questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Drummond, PhD, Study Director — University of Calgary
Locations (1):
- Alberta Health Services Chronic Pain Centre, Calgary, Alberta, Canada